CLINICAL TRIAL: NCT01830244
Title: Tailored Neoadjuvant Epirubicin and Cyclophosphamide (EC) and Nanoparticle Albumin Bound (Nab) Paclitaxel for Newly Diagnosed Breast Cancer
Brief Title: IST Neoadjuvant Abraxane in Newly Diagnosed Breast Cancer
Acronym: Neonab
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Barwon Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALCC12.01
Record Dates: First submitted 2013-03-27; First posted 2013-04-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: chemotherapy; nab paclitaxel; neoadjuvant therapy; breast cancer; pathologic complete response
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nab-Paclitaxel 125mg/m2 (Experimental): Epirubicin 90 mg/m2 and cyclophosphamide 600mg/m2 IV every 3 weeks for 4 cycles.
  Nab paclitaxel 125mg/m2 IV days 1, 8 and 15 for 12 weeks In case of HER2 positive tumour patients will receive trastuzumab in combination with nab-Paclitaxel
  Interventions: Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Nab-Paclitaxel — Nab-Paclitaxel- 125 mg/m2 days 1,8, 15 for 12 weeks
  Other Names: Abraxane

SUMMARY:
The aim of this project is to evaluate tailored primary systemic therapy with sequential nab paclitaxel and epirubicin and cyclophosphamide in early breast cancer. This study will be an open label phase II clinical trial. The hypothesis is that tailored neoadjuvant chemotherapy with sequential nab paclitaxel and epirubicin and cyclophosphamide is feasible and achieves high response rates. It is proposed that 60 patients will be enrolled in this study including 40 patients which are likely to have chemotherapy sensitive tumors and 20 patients who have ER positive tumors and are more likely to respond to hormonal treatment as an exploratory cohort. The target population is women with early breast cancer who are eligible for primary systemic therapy. The overall response rate in the breast will be measured. Secondary endpoints will include response rates in axillary lymph nodes, safety and tolerability and the rate of breast conservation. Participants will have a blood test to determine a specific genotype status that may help in predicting sensitivity to chemotherapy. This genotype test result is exploratory and will not influence selection of therapy for participants. Patients will also be given the option of having he their tumour tissues used in laboratory studies involving isolating cancer initiating cells from the tumor to subsequently generate breast cancer models in the laboratory and using aptamers (chemical antibodies) to target tumours.

DETAILED DESCRIPTION:
The prognosis and survival rate of breast cancer varies depending on the extent of the disease, performance status of patients and the type of tumour including the status of oestrogen receptor (ER), progesterone receptor (PR) and human epidermal growth factor receptor 2 (HER2). Expression of ER and PR generally indicates better prognosis than the overexpression of HER2 and triple negative breast cancer generally indicates more aggressive cancers with a high growth rate [1].

Preoperative or neoadjuvant therapy which is also known as primary systemic therapy followed by surgery and adjuvant radiation therapy is recommended for patients with locally advanced breast cancer [2]. Studies using primary systemic therapy have demonstrated useful rates of clinical response and pathological complete response(pCR) rates in the breast alone and pathological complete response rates in the axillary notes. The response rates vary considerably, however response rates to cytotoxic chemotherapy have been uniformally higher in ER negative tumors. There is additional improvement in the pathological complete response rates of about 10 % with the addition of a taxane [4]. For operable breast cancer, primary systemic therapy can be considered as an alternative to adjuvant systemic therapy for patients who require a mastectomy but who desire breast conservation surgery. In patients with large tumours who can technically have a lumpectomy, primary systemic therapy may permit less extensive surgery and may result in a better cosmetic result. Primary systemic therapy may also be advisable in patients who have medical contraindications to surgery or where delayed surgery is required.

Nanoparticle albumin bound paclitaxel is reported to achieve a higher intracellular tumour paclitaxel concentration via the albumin mediated transendothelial transport system [5]. Better tolerability and efficacy has been demonstrated when compared to paclitaxel or docetaxel in the treatment of metastatic breast cancer [6, 7]. Nab paclitaxel is being evaluated in the adjuvant treatment of patients with breast cancer [8, 9] and in the neoadjuvant setting [10.] The preoperative setting provides an opportunity to study the early molecular changes that may occur in response to treatment. Alteration of biomarkers between pre and post chemotherapy including hormone receptors, the Human Epidermal growth factor receptor (HER2)and Ki67 [11, 12] as well as gene pathways [13] are areas of possible exploration in neoadjuvant studies whereby tissue is available for analysis before and after the chemotherapy treatment. Particular patterns of reduction in tumour size on MRI can be predictive of successful response, detecting residual tumour not apparent on mammogram or U/S and in accurate evaluation of tumour volume [14.] Functional imaging biomarkers of response also have potential utility in assessing treatment response [15.] A recent study reported that 4 cycles of adjuvant therapy with the combination of nab Paclitaxel and cyclophosphamide, with or without trastuzumab, is feasible and well tolerated in patients with early stage breast cancer. Another small study demonstrated feasibility of nab Paclitaxel followed by 5-fluorouracil, epirubicin and cyclophosphamide (FEC) [16.] An anthracycline containing regimen followed by conventional paclitaxel is amongst the most commonly prescribed adjuvant chemotherapy regime for early breast cancer. Cyclophosphamide is given in combination with doxorubicin or its epimer epirubicin. Epirubicin achieves similar efficacy results to doxorubicin but causes less cardiotoxicity [17 19].

Although standards of care are varied, adjuvant chemotherapy in 2011 is generally recommended in women with triple negative breast cancer (TNBC) and HER amplified tumors. In women with hormone receptor positive tumors without HER2 amplification, chemotherapy is reserved for tumors that are large or with extensive nodal involvement and/ or high risk biology. The latter includes young age, presence of lymphovascular space invasion, a high proliferative index (Ki67 expression), lower ER/PR expression, higher Oncotype Dx score and luminal B tumors[20]. Thus there are evolving trends to tailor therapy based on the tumor characteristics indicating perceived risk, patient factors, particularly comorbid illness and patient preferences as well as prediction of response.

In breast cancer, immunohistochemical assessment of the proportion of cells staining for the nuclear antigen Ki67 has become a widely used method for comparing proliferation between tumour samples[21]. Potential uses include prognosis, prediction of relative responsiveness or resistance to chemotherapy or endocrine therapy, estimation of residual risk in patients on standard therapy and as a dynamic biomarker of treatment efficacy in samples taken before, during, and after neoadjuvant therapy[21, 22]. Ki67 labeling Index has been incorporated as one of the means of identifying tumor subtypes by the 2011 St Gallen International Expert Consensus on the Primary Therapy of Early Breast Cancer[20]. Analysis of gene expression arrays has resulted in the recognition of several fundamentally different subtypes of breast cancer[23]. Using gene expression profile distinction can be made between luminal A and luminal B tumors. While both subtypes could be ER positive but luminal A tumours are unlikely to benefit from cytotoxic chemotherapy. Because it is not always feasible to obtain gene expression array information, a simplified classification, closely following that proposed by Cheang et al whereby a cutpoint for Ki67 labeling index of <15% was established by comparison with PAM50 intrinsic subtyping to differentiate between luminal A and luminal B tumours[24]. Local quality control of Ki67 staining is important[20].

The Oncotype Recurrence Score is a validated a 21-gene assay that is now offered as a commercial reference laboratory test (Oncotype DX, Genomic Health Inc. Redwood City, CA). The 21-gene panel includes genes involved in tumour cell proliferation and hormonal response, characteristics that have been reported to be associated with chemotherapy response in general. Oncotype DX not only quantifies the likelihood of breast cancer recurrence in women with node-negative, oestrogen receptor-positive breast cancer, but also predicts the magnitude of chemotherapy benefit [21, 26]. Likelihood of chemotherapy benefit is reported as low (Recurrence Score <18, intermediate RS 18-30 and high >30).[26] The main utility of Oncotype DX is in the adjuvant setting where it could be a powerful tool to guide decision regarding the role of cytotoxic chemotherapy in hormone positive tumours. In this neoadjuvant study we will employ Oncotype DX to guide decision about use of chemotherapy in patients with tumours that have high Ki67 (>15) but low ER expression and also in the other groups that may have low Ki67 (<15) but high ER expression by IHC.

The goal is to use the best combination, sequence and duration of therapy together with predicting and monitoring response with high fidelity in the individual patient. Further studies are needed to optimize treatment regimens so as to increase pathologic response rates and ultimately survival, with a further goal of reducing risk and adverse events.

This study uses a tailored approach to select treatment involving the choice of NAB Paclitaxel and EC based on the individual patient and tumour characteristics.

Breast Cancer Stem Cells

It is now widely accepted that our inability to cure cancer is largely due to the presence of a subset of cells within a cancer that constitutes a reservoir of self sustaining [25]. Current radiation and cytotoxic chemotherapies more effectively destroy the proliferating cells that form the bulk of the tumour, but are largely ineffective against the cancer stem cells (CSC)[26, 27]. Breast cancer was the first solid malignancy from which CSCs were identified[28], via specific cell surface marker proteins CD44 and epithelial cell adhesion molecules (EpCAM)[29, 30]. EpCAM and CD44v6 are among best available, clinically relevant breast cancer stem cell markers for the proof of principle work in this project [30] .

Aptamers

Aptamers are short, singlestranded RNA or DNA that fold into specific 3D structures and bind to their target molecules with high affinity and specificity[31]. Unlike antibodies, aptamers remain structurally stable across a wide range of temperature and storage conditions. They are generally nonimmunogenic, nontoxic and are 20 to 25 times smaller than monoclonal antibodies. Thus aptamers offer several advantages for tissue penetration and have shorter circulation time and faster body clearance resulting in a low background noise during imaging and lower radiation dose. In addition, aptamers can be produced rapidly, relatively inexpensively, and with high homogeneity [32, 33].

HDACi

Histone deacetylases (HDACs) play an important role in gene regulation. Inhibitors of HDACs (HDACi) are novel anticancer drugs, which induce histone (hyper) acetylation and counteract aberrant gene repression[34]. HDACi also evoke nonhistone protein acetylation, which can alter signalling networks relevant for tumorigenesis and these agents can also promote the degradation of (proto) oncoproteins. Adult stem cells are maintained in a quiescent state but are able to exit quiescence and rapidly expand and differentiate in response to stress. The quiescence of cancer stem cells (CSCs) is highly relevant to cancer therapy since the quiescent CSC is often resistant to both conventional therapy and targeted therapies. The p53 gene plays a critical role in regulating stem cell quiescence [35]. CSCs promote chemotherapy and radiation resistance through an increase in DNA repair capacity and in histone H3 deacetylation[35]. Recently the role of HDACi in moving latent or quiescent cells to an activated state and sensitizing them to other treatments has become a focus of investigation in both HIV and cancer. The HDAC inhibitors have been studied in many hematologic and solid malignancies but little work has focused on breast cancer and particularly CSC[36, 37]. A study of HDACi on quiescent CSCs in breast tumours and their radiation and chemotherapy responses would be of great interest in developing new therapeutic paradigms using this class of agents.

NAD(P)H:quinone oxidoreductase 1 and NQO1*2 genotype (P187S)

Nicotinamide adenine dinucleotide, (NAD+), is a coenzyme found in all cells. In metabolism, NAD+ is involved in reduction oxidation (redox) reactions, carrying electrons from one reaction to another. The coenzyme is found as NAD+, which is an oxidizing agent and forms NADH. This can then be used as a reducing agent. Electron transfer reactions are the main function of NAD+. However, it is also used in other cellular processes, the most notable one being a substrate of enzymes that add or remove chemical groups from proteins, in posttranslational modifications. There is evidence that genetic variants in oxidative stress related genes predict resistance to chemotherapy in primary breast cancer and that germline polymorphisms can affect chemotherapy sensitivity in patients with breastcancer[38].

The status of superoxide dismutases and NAD (P) H quinone oxidoreductases have prognostic significance in breast carcinomas[39]. The NQO1 enzyme guards against oxidative stress and carcinogenesis and stabilizes p53 tumor suppressor[40, 41]. NQO1 deficient mice show reduced p53 induction and apoptosis. NQO1*2 is a missense variant (NP_000894:p.187P4S) that is homozygous in 4-20% of human population[42]. Cells with the homozygous NQO1*2 genotype have no measurable NQO1 activity, reflecting the very low levels of the NQO1 P187S protein, which undergoes rapid turnover via the ubiquitin proteasome pathway[43]. Response to epirubicin is impaired in NQO1*2homozygous breast carcinoma cells in vitro, reflecting both p53linked and p53independentroles of NQO1. A potential defective anthracycline response in NQO1deficient breast tumors may confer increased genomic instability promoted by elevated reactive oxygen species, and suggest that the NQO1 genotype is a prognostic and predictive marker for breast cancer. A homozygous common missense variant (NQO1*2, rs1800566(T), NM_000903.2:c.558C4T) that disables NQO1 strongly has been shown to predicts poor survival among two independent series of women with breast cancer, an effect particularly evident after anthracycline based adjuvant chemotherapy with epirubicin[44]. As part of this study the NQO1*2 genotype status of all patients will be assessed. A correlation can be explored between NQO1*2 genotype status and response rate in this setting. The study will evaluate the feasibility and safety of tailored primary systemic therapy in the study population.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have consented to participate and must have signed and dated an appropriate approved consent form.
* Female 18 Years and older
* The Eastern Cooperative Oncology Group (ECOG) performance status must be 0 or 1
* The diagnosis of invasive adenocarcinoma of the breast must have been made by core needle biopsy or limited incisional biopsy.
* Patients must have tumor diameter >2 cm measurable at least clinically; by physical exam, unless the patient has inflammatory breast cancer, in which case measurable disease by physical exam is not required or ultrasonographic staging (T2, T3 or T4 a, b, c tumours with any clinical node status N0-N2).
* Left ventricular ejection fraction (LVEF) assessment by 2-D echocardiogram or Multi Gated Acquisition Scan (MUGA scan) performed within 3 months prior to study entry must be greater or equal to 50%.
* Adequate haematological, renal and hepatic function (neutrophils >=2 × 109/L, platelets ≥100 × 109/L, hemoglobin >=100g/L, total bilirubin ≤ 1.5 upper limit of normal (ULN), aspartate aminotransferase and alanine aminotransferase ≤1.5 × ULN, alkaline phosphatases ≤2.5 ULN, creatinine ≤ 1.5 ULN).
* Negative pregnancy test

Exclusion Criteria:

* Severe cardiovascular, hepatic, neurologic or renal comorbid conditions
* Primary surgical treatment of the tumor or excisional biopsy or lumpectomy performed prior to study entry.
* Surgical axillary staging procedure prior to study entry.
* Definitive clinical or radiologic evidence of metastatic disease.
* History of ipsilateral invasive breast cancer regardless of treatment or ipsilateral ductal carcinoma in situ (DCIS) treated with radiotherapy (RT).
* Non-breast malignancies unless the patient is considered to be disease-free for 5 or more years prior to study entry and is deemed by her physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Previous therapy with anthracyclines or taxanes for any malignancy.
* Treatment including RT, chemotherapy, and/or targeted therapy, administered for the currently diagnosed breast cancer prior to study entry.
* Continued therapy with any hormonal agent such as raloxifene, tamoxifen, or other Selective estrogen receptor modulator (SERM).
* Any sex hormonal therapy, e.g., birth control pills and ovarian hormone replacement therapy
* History of hepatitis B or C.
* Sensory/motor neuropathy greater or equal to grade 2, as defined by the current version of the NCI's CTCAE.
* Pregnancy or continuing lactation at the time of study entry.
* Use of any investigational agent within 4 weeks prior to enrollment in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-09 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response in the breast | 24 weeks (time window + 4 weeks)
  Pathological complete response defined as breast only, ypT0/ ypTis regardless of nodal status

SECONDARY OUTCOMES:
Pathologic Response rate in breast and axillary lymph nodes | 24 weeks (time window + 4 weeks)
  Pathologic assessment
Rate of pathologic complete response and near complete response in the breast combined | 24 weeks (time window + 4 weeks)
  Pathologic assessment
Breast conservation rate | 24 weeks (time window + 4 weeks)
Progression Free Survival | 5 years
Safety and tolerability | During treatment (24 weeks)
  Safety will be measured using NCI Common Toxicity Criteria for Adverse Effects version 4.0

OTHER OUTCOMES:
NQ01*2 genotype (P187S) status | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Khasraw, MD, Principal Investigator — Barwon Health
Locations (5):
- Australia (5):
  - Bankstown Lidcome Hospital, Bankstown, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Barwon Health, Geelong, Victoria
  - St John of God Healthcare, Geelong, Geelong, Victoria
  - South West Healthcare, Warrnambool, Victoria

REFERENCES:
- [Background] Foulkes WD, Smith IE, Reis-Filho JS. Triple-negative breast cancer. N Engl J Med. 2010 Nov 11;363(20):1938-48. doi: 10.1056/NEJMra1001389. PMID 21067385
- [Background] Kaufmann M, Hortobagyi GN, Goldhirsch A, Scholl S, Makris A, Valagussa P, Blohmer JU, Eiermann W, Jackesz R, Jonat W, Lebeau A, Loibl S, Miller W, Seeber S, Semiglazov V, Smith R, Souchon R, Stearns V, Untch M, von Minckwitz G. Recommendations from an international expert panel on the use of neoadjuvant (primary) systemic treatment of operable breast cancer: an update. J Clin Oncol. 2006 Apr 20;24(12):1940-9. doi: 10.1200/JCO.2005.02.6187. PMID 16622270
- [Background] Bear HD, Anderson S, Brown A, Smith R, Mamounas EP, Fisher B, Margolese R, Theoret H, Soran A, Wickerham DL, Wolmark N; National Surgical Adjuvant Breast and Bowel Project Protocol B-27. The effect on tumor response of adding sequential preoperative docetaxel to preoperative doxorubicin and cyclophosphamide: preliminary results from National Surgical Adjuvant Breast and Bowel Project Protocol B-27. J Clin Oncol. 2003 Nov 15;21(22):4165-74. doi: 10.1200/JCO.2003.12.005. Epub 2003 Oct 14. PMID 14559892
- [Background] Gradishar WJ, Wedam SB, Jahanzeb M, Erban J, Limentani SA, Tsai KT, Olsen SR, Swain SM. Neoadjuvant docetaxel followed by adjuvant doxorubicin and cyclophosphamide in patients with stage III breast cancer. Ann Oncol. 2005 Aug;16(8):1297-304. doi: 10.1093/annonc/mdi254. Epub 2005 May 19. PMID 15905305
- [Background] Foote M. Using nanotechnology to improve the characteristics of antineoplastic drugs: improved characteristics of nab-paclitaxel compared with solvent-based paclitaxel. Biotechnol Annu Rev. 2007;13:345-57. doi: 10.1016/S1387-2656(07)13012-X. PMID 17875482
- [Background] Gradishar WJ, Krasnojon D, Cheporov S, Makhson AN, Manikhas GM, Clawson A, Bhar P. Significantly longer progression-free survival with nab-paclitaxel compared with docetaxel as first-line therapy for metastatic breast cancer. J Clin Oncol. 2009 Aug 1;27(22):3611-9. doi: 10.1200/JCO.2008.18.5397. Epub 2009 May 26. PMID 19470941
- [Background] Gradishar WJ, Tjulandin S, Davidson N, Shaw H, Desai N, Bhar P, Hawkins M, O'Shaughnessy J. Phase III trial of nanoparticle albumin-bound paclitaxel compared with polyethylated castor oil-based paclitaxel in women with breast cancer. J Clin Oncol. 2005 Nov 1;23(31):7794-803. doi: 10.1200/JCO.2005.04.937. Epub 2005 Sep 19. PMID 16172456
- [Background] Yardley D, Burris H 3rd, Peacock N, Raefsky E, Melnik M, Inhorn R, Shipley D, Hainsworth J. A pilot study of adjuvant nanoparticle albumin-bound (nab) paclitaxel and cyclophosphamide, with trastuzumab in HER2-positive patients, in the treatment of early-stage breast cancer. Breast Cancer Res Treat. 2010 Sep;123(2):471-5. doi: 10.1007/s10549-010-1047-0. Epub 2010 Jul 24. PMID 20658263
- [Background] Dang C, Fornier M, Sugarman S, Troso-Sandoval T, Lake D, D'Andrea G, Seidman A, Sklarin N, Dickler M, Currie V, Gilewski T, Moynahan ME, Drullinsky P, Robson M, Wasserheit-Leiblich C, Mills N, Steingart R, Panageas K, Norton L, Hudis C. The safety of dose-dense doxorubicin and cyclophosphamide followed by paclitaxel with trastuzumab in HER-2/neu overexpressed/amplified breast cancer. J Clin Oncol. 2008 Mar 10;26(8):1216-22. doi: 10.1200/JCO.2007.12.0733. PMID 18323546
- [Background] Kaklamani VG, Siziopikou K, Scholtens D, Lacouture M, Gordon J, Uthe R, Meservey C, Hansen N, Khan SA, Jeruss JS, Bethke K, Cianfrocca M, Rosen S, Von Roenn J, Wayne J, Parimi V, Jovanovic B, Gradishar W. Pilot neoadjuvant trial in HER2 positive breast cancer with combination of nab-paclitaxel and lapatinib. Breast Cancer Res Treat. 2012 Apr;132(3):833-42. doi: 10.1007/s10549-011-1411-8. Epub 2011 Feb 27. PMID 21359953
- [Background] Khasraw M, Brogi E, Seidman AD. The need to examine metastatic tissue at the time of progression of breast cancer: is re-biopsy a necessity or a luxury? Curr Oncol Rep. 2011 Feb;13(1):17-25. doi: 10.1007/s11912-010-0137-9. PMID 21053108
- [Background] Kumaki N, Umemura S, Tang X, Saito Y, Suzuki Y, Tokuda Y. Alteration of immunohistochemical biomarkers between pre- and post-chemotherapy: hormone receptors, HER2 and Ki-67. Breast Cancer. 2011 Apr;18(2):98-102. doi: 10.1007/s12282-010-0238-1. Epub 2011 Feb 3. PMID 21290265
- [Background] Iwamoto T, Bianchini G, Booser D, Qi Y, Coutant C, Shiang CY, Santarpia L, Matsuoka J, Hortobagyi GN, Symmans WF, Holmes FA, O'Shaughnessy J, Hellerstedt B, Pippen J, Andre F, Simon R, Pusztai L. Gene pathways associated with prognosis and chemotherapy sensitivity in molecular subtypes of breast cancer. J Natl Cancer Inst. 2011 Feb 2;103(3):264-72. doi: 10.1093/jnci/djq524. Epub 2010 Dec 29. PMID 21191116
- [Background] Partridge SC, Gibbs JE, Lu Y, Esserman LJ, Tripathy D, Wolverton DS, Rugo HS, Hwang ES, Ewing CA, Hylton NM. MRI measurements of breast tumor volume predict response to neoadjuvant chemotherapy and recurrence-free survival. AJR Am J Roentgenol. 2005 Jun;184(6):1774-81. doi: 10.2214/ajr.184.6.01841774. PMID 15908529
- [Background] O'Flynn EA, DeSouza NM. Functional magnetic resonance: biomarkers of response in breast cancer. Breast Cancer Res. 2011 Feb 23;13(1):204. doi: 10.1186/bcr2815. PMID 21392409
- [Background] Robidoux A, Buzdar AU, Quinaux E, Jacobs S, Rastogi P, Fourchotte V, Younan RJ, Pajon ER, Shalaby IA, Desai AM, Fehrenbacher L, Geyer CE Jr, Mamounas EP, Wolmark N. A phase II neoadjuvant trial of sequential nanoparticle albumin-bound paclitaxel followed by 5-fluorouracil/epirubicin/cyclophosphamide in locally advanced breast cancer. Clin Breast Cancer. 2010 Feb;10(1):81-6. doi: 10.3816/CBC.2010.n.011. PMID 20133263
- [Background] Findlay B, Tonkin K, Crump M, Norris B, Trudeau M, Blackstein M, Burnell M, Skillings J, Bowman D, Walde D, Levine M, Pritchard KI, Palmer MJ, Tu D, Shepherd L. A dose escalation trial of adjuvant cyclophosphamide and epirubicin in combination with 5-fluorouracil using G-CSF support for premenopausal women with breast cancer involving four or more positive nodes. Ann Oncol. 2007 Oct;18(10):1646-51. doi: 10.1093/annonc/mdm277. Epub 2007 Aug 22. PMID 17716984
- [Background] Khasraw M, Bell R, Dang C. Epirubicin: is it like doxorubicin in breast cancer? A clinical review. Breast. 2012 Apr;21(2):142-9. doi: 10.1016/j.breast.2011.12.012. Epub 2012 Jan 17. PMID 22260846
- [Background] Goldhirsch A, Wood WC, Coates AS, Gelber RD, Thurlimann B, Senn HJ; Panel members. Strategies for subtypes--dealing with the diversity of breast cancer: highlights of the St. Gallen International Expert Consensus on the Primary Therapy of Early Breast Cancer 2011. Ann Oncol. 2011 Aug;22(8):1736-47. doi: 10.1093/annonc/mdr304. Epub 2011 Jun 27. PMID 21709140
- [Background] Dowsett M, Nielsen TO, A'Hern R, Bartlett J, Coombes RC, Cuzick J, Ellis M, Henry NL, Hugh JC, Lively T, McShane L, Paik S, Penault-Llorca F, Prudkin L, Regan M, Salter J, Sotiriou C, Smith IE, Viale G, Zujewski JA, Hayes DF; International Ki-67 in Breast Cancer Working Group. Assessment of Ki67 in breast cancer: recommendations from the International Ki67 in Breast Cancer working group. J Natl Cancer Inst. 2011 Nov 16;103(22):1656-64. doi: 10.1093/jnci/djr393. Epub 2011 Sep 29. PMID 21960707
- [Background] Untch M, Loibl S, Konecny GE, von Minckwitz G. Neoadjuvant clinical trials for the treatment of primary breast cancer: the experience of the German study groups. Curr Oncol Rep. 2012 Feb;14(1):27-34. doi: 10.1007/s11912-011-0212-x. PMID 22246608
- [Background] Perou CM, Sorlie T, Eisen MB, van de Rijn M, Jeffrey SS, Rees CA, Pollack JR, Ross DT, Johnsen H, Akslen LA, Fluge O, Pergamenschikov A, Williams C, Zhu SX, Lonning PE, Borresen-Dale AL, Brown PO, Botstein D. Molecular portraits of human breast tumours. Nature. 2000 Aug 17;406(6797):747-52. doi: 10.1038/35021093. PMID 10963602
- [Background] Cheang MC, Chia SK, Voduc D, Gao D, Leung S, Snider J, Watson M, Davies S, Bernard PS, Parker JS, Perou CM, Ellis MJ, Nielsen TO. Ki67 index, HER2 status, and prognosis of patients with luminal B breast cancer. J Natl Cancer Inst. 2009 May 20;101(10):736-50. doi: 10.1093/jnci/djp082. Epub 2009 May 12. PMID 19436038
- [Background] Visvader JE. Cells of origin in cancer. Nature. 2011 Jan 20;469(7330):314-22. doi: 10.1038/nature09781. PMID 21248838
- [Background] Zoller M. CD44: can a cancer-initiating cell profit from an abundantly expressed molecule? Nat Rev Cancer. 2011 Apr;11(4):254-67. doi: 10.1038/nrc3023. Epub 2011 Mar 10. PMID 21390059
- [Background] Al-Hajj M, Wicha MS, Benito-Hernandez A, Morrison SJ, Clarke MF. Prospective identification of tumorigenic breast cancer cells. Proc Natl Acad Sci U S A. 2003 Apr 1;100(7):3983-8. doi: 10.1073/pnas.0530291100. Epub 2003 Mar 10. PMID 12629218
- [Background] Stratford AL, Reipas K, Maxwell C, Dunn SE. Targeting tumour-initiating cells to improve the cure rates for triple-negative breast cancer. Expert Rev Mol Med. 2010 Jul 26;12:e22. doi: 10.1017/S1462399410001535. PMID 20653987
- [Background] Hebbard L, Steffen A, Zawadzki V, Fieber C, Howells N, Moll J, Ponta H, Hofmann M, Sleeman J. CD44 expression and regulation during mammary gland development and function. J Cell Sci. 2000 Jul;113 ( Pt 14):2619-30. doi: 10.1242/jcs.113.14.2619. PMID 10862719
- [Background] Munz M, Baeuerle PA, Gires O. The emerging role of EpCAM in cancer and stem cell signaling. Cancer Res. 2009 Jul 15;69(14):5627-9. doi: 10.1158/0008-5472.CAN-09-0654. Epub 2009 Jul 7. PMID 19584271
- [Background] Shigdar S, Ward AC, De A, Yang CJ, Wei M, Duan W. Clinical applications of aptamers and nucleic acid therapeutics in haematological malignancies. Br J Haematol. 2011 Oct;155(1):3-13. doi: 10.1111/j.1365-2141.2011.08807.x. Epub 2011 Aug 2. PMID 21810089
- [Background] Yu C, Hu Y, Duan J, Yuan W, Wang C, Xu H, Yang XD. Novel aptamer-nanoparticle bioconjugates enhances delivery of anticancer drug to MUC1-positive cancer cells in vitro. PLoS One. 2011;6(9):e24077. doi: 10.1371/journal.pone.0024077. Epub 2011 Sep 1. PMID 21912664
- [Background] Wu S, Duan N, Wang Z, Wang H. Aptamer-functionalized magnetic nanoparticle-based bioassay for the detection of ochratoxin A using upconversion nanoparticles as labels. Analyst. 2011 Jun 7;136(11):2306-14. doi: 10.1039/c0an00735h. Epub 2011 Apr 8. PMID 21479303
- [Background] Buchwald M, Kramer OH, Heinzel T. HDACi--targets beyond chromatin. Cancer Lett. 2009 Aug 8;280(2):160-7. doi: 10.1016/j.canlet.2009.02.028. Epub 2009 Apr 1. PMID 19342155
- [Background] Li L, Bhatia R. Stem cell quiescence. Clin Cancer Res. 2011 Aug 1;17(15):4936-41. doi: 10.1158/1078-0432.CCR-10-1499. Epub 2011 May 18. PMID 21593194
- [Background] Tan J, Cang S, Ma Y, Petrillo RL, Liu D. Novel histone deacetylase inhibitors in clinical trials as anti-cancer agents. J Hematol Oncol. 2010 Feb 4;3:5. doi: 10.1186/1756-8722-3-5. PMID 20132536
- [Background] Lemoine M, Younes A. Histone deacetylase inhibitors in the treatment of lymphoma. Discov Med. 2010 Nov;10(54):462-70. PMID 21122478
- [Background] Yu KD, Huang AJ, Fan L, Li WF, Shao ZM. Genetic variants in oxidative stress-related genes predict chemoresistance in primary breast cancer: a prospective observational study and validation. Cancer Res. 2012 Jan 15;72(2):408-19. doi: 10.1158/0008-5472.CAN-11-2998. Epub 2011 Dec 6. PMID 22147260
- [Background] Hubackova M, Vaclavikova R, Ehrlichova M, Mrhalova M, Kodet R, Kubackova K, Vrana D, Gut I, Soucek P. Association of superoxide dismutases and NAD(P)H quinone oxidoreductases with prognosis of patients with breast carcinomas. Int J Cancer. 2012 Jan 15;130(2):338-48. doi: 10.1002/ijc.26006. Epub 2011 Apr 20. PMID 21351093
- [Background] Anwar A, Dehn D, Siegel D, Kepa JK, Tang LJ, Pietenpol JA, Ross D. Interaction of human NAD(P)H:quinone oxidoreductase 1 (NQO1) with the tumor suppressor protein p53 in cells and cell-free systems. J Biol Chem. 2003 Mar 21;278(12):10368-73. doi: 10.1074/jbc.M211981200. Epub 2003 Jan 14. PMID 12529318
- [Background] Tsvetkov P, Reuven N, Shaul Y. Ubiquitin-independent p53 proteasomal degradation. Cell Death Differ. 2010 Jan;17(1):103-8. doi: 10.1038/cdd.2009.67. PMID 19557012
- [Background] Nioi P, Hayes JD. Contribution of NAD(P)H:quinone oxidoreductase 1 to protection against carcinogenesis, and regulation of its gene by the Nrf2 basic-region leucine zipper and the arylhydrocarbon receptor basic helix-loop-helix transcription factors. Mutat Res. 2004 Nov 2;555(1-2):149-71. doi: 10.1016/j.mrfmmm.2004.05.023. PMID 15476858
- [Background] Siegel D, Anwar A, Winski SL, Kepa JK, Zolman KL, Ross D. Rapid polyubiquitination and proteasomal degradation of a mutant form of NAD(P)H:quinone oxidoreductase 1. Mol Pharmacol. 2001 Feb;59(2):263-8. doi: 10.1124/mol.59.2.263. PMID 11160862
- [Background] Fagerholm R, Hofstetter B, Tommiska J, Aaltonen K, Vrtel R, Syrjakoski K, Kallioniemi A, Kilpivaara O, Mannermaa A, Kosma VM, Uusitupa M, Eskelinen M, Kataja V, Aittomaki K, von Smitten K, Heikkila P, Lukas J, Holli K, Bartkova J, Blomqvist C, Bartek J, Nevanlinna H. NAD(P)H:quinone oxidoreductase 1 NQO1*2 genotype (P187S) is a strong prognostic and predictive factor in breast cancer. Nat Genet. 2008 Jul;40(7):844-53. doi: 10.1038/ng.155. Epub 2008 May 30. PMID 18511948
- [Derived] Murphy C, Muscat A, Ashley D, Mukaro V, West L, Liao Y, Chisanga D, Shi W, Collins I, Baron-Hay S, Patil S, Lindeman G, Khasraw M. Tailored NEOadjuvant epirubicin, cyclophosphamide and Nanoparticle Albumin-Bound paclitaxel for breast cancer: The phase II NEONAB trial-Clinical outcomes and molecular determinants of response. PLoS One. 2019 Feb 14;14(2):e0210891. doi: 10.1371/journal.pone.0210891. eCollection 2019. PMID 30763338
- [Derived] Murphy C, Mukaro V, Tobler R, Asher R, Gibbs E, West L, Giuffre B, Baron-Hay S, Khasraw M. Evaluating the role of magnetic resonance imaging post-neoadjuvant therapy for breast cancer in the NEONAB trial. Intern Med J. 2018 Jun;48(6):699-705. doi: 10.1111/imj.13617. PMID 28869790